CLINICAL TRIAL: NCT00681850
Title: OPtimal Type 2 dIabetes Management Including Benchmarking and Standard trEatment.
Acronym: Optimise
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Eugène Vissers, MD, Therapeutic Area Leader Cardivascular and Diabetes., AstraZeneca Pharmaceuticals
Other Study IDs: D3560L00071
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2010-06

CONDITIONS: Diabetes
Keywords: Diabetes; Benchmarking; quality of patient care; Diabetic Population
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Control group
- 2: Benchmarking group

SUMMARY:
Demonstrate that the use of benchmarking improves quality of patient care, in particular the control of diabetes, lipids and blood pressure, by determining the percentage of patients in the benchmarking group achieving pre-set targets for HbA1c 14,18, LDL-cholesterol16,18 and Systolic Blood Pressure17,18 versus control group (non-benchmarking group) after 12 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed Consent
* Patients suffering from diabetes type II, insulin dependent or not insulin dependent.

Exclusion Criteria:

* Type I diabetes
* Pregnancy diabetes
* Hospitalisation, as this is a primary care study
* Patients who are member of the Belgian Diabetes Convention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General Practioners
Sampling Method: Probability Sample
Enrollment: 4027 (Actual)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
HbA1c, LDL-cholesterol, Systolic Blood Pressure | Visit 1; Visit 2 (after approximately 4 months after visit 1); Visit 3 (after approximately 8 months after visit 1); Visit 4 (after approximately 12 months after visit 1)

SECONDARY OUTCOMES:
Glycaemia, Triglycerides, Total and HDL-Cholesterol, Diastolic Blood Pressure, Waist circumference, Smoking habits, Microalbuminuria, Body Mass Index, Physical activity (Rating scale and step counter), Degree of ophthalmic control and dietary advice | Visit 1Visit 2 (after approximately 4 months after visit 1)Visit 3 (after approximately 8 months after visit 1)Visit 4 (after approximately 12 months after visit 1)

CONTACTS AND LOCATIONS:
Overall Officials: Hermans, M. Prof., Principal Investigator — UCL
Locations (252):
- Belgium (150):
  - Research Site, Aalst
  - Research Site, Aarschot
  - Research Site, Alsemberg
  - Research Site, Amay
  - Research Site, Antoing
  - Research Site, Antwerp
  - Research Site, Anzegem
  - Research Site, Ath
  - Research Site, Baisy-Thy
  - Research Site, Balleul
  - Research Site, Bastogne
  - Research Site, Battice
  - Research Site, Beerse
  - Research Site, Bellaire
  - Research Site, Bertogne
  - Research Site, Betekom
  - Research Site, Beveren
  - Research Site, Bilzen
  - Research Site, Binche
  - Research Site, Boezinge
  - Research Site, Boirs
  - Research Site, Borgerhout
  - Research Site, Bouillon
  - Research Site, Brain-l'alleud
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Cercxhe-heuseux
  - Research Site, Champion
  - Research Site, Clabeoq
  - Research Site, Corbion
  - Research Site, De Pinte
  - Research Site, Diest
  - Research Site, Dottignies
  - Research Site, Dworp
  - Research Site, Ekeren
  - Research Site, Enghien
  - Research Site, Erembodegem
  - Research Site, Essen
  - Research Site, Eupen
  - Research Site, Geel
  - Research Site, Genk
  - Research Site, Genly
  - Research Site, Geraardsbergen
  - Research Site, Ghent
  - Research Site, Ghlin
  - Research Site, Gilly
  - Research Site, Gozée
  - Research Site, Gribomont
  - Research Site, Haaltert
  - Research Site, Halen
  - Research Site, Halle
  - Research Site, Ham
  - Research Site, Hannut
  - Research Site, Hasselt
  - Research Site, Havinnes
  - Research Site, Havré
  - Research Site, Herent
  - Research Site, Herstal
  - Research Site, Herzele
  - Research Site, Hoboken
  - Research Site, Hooglede
  - Research Site, Houthalen-Helchteren
  - Research Site, Incourt
  - Research Site, Jemappes
  - Research Site, Kapellen
  - Research Site, Knokke
  - Research Site, Kuringen
  - Research Site, La Hulpe
  - Research Site, La Louvière
  - Research Site, La Roche
  - Research Site, Laakdal
  - Research Site, Lanaken
  - Research Site, Lauwe
  - Research Site, Lessines
  - Research Site, Libramont
  - Research Site, Lier
  - Research Site, Liège
  - Research Site, Ligne
  - Research Site, Ligney
  - Research Site, Linkebeek
  - Research Site, Lo-reninge
  - Research Site, Louveigné
  - Research Site, Manage
  - Research Site, Marche
  - Research Site, Marchin
  - Research Site, Marchovelette
  - Research Site, Marloie
  - Research Site, Mechelen
  - Research Site, Merksem
  - Research Site, Merksplas
  - Research Site, Mettet
  - Research Site, Moerkerke
  - Research Site, Mol
  - Research Site, Moorlede
  - Research Site, Moorsel
  - Research Site, Mouscron
  - Research Site, Noorderwijk
  - Research Site, Olen
  - Research Site, Ooigem
  - Research Site, Oostrozebeke
  - Research Site, Oppuurs
  - Research Site, Ostend
  - Research Site, Outer
  - Research Site, Perk
  - Research Site, Pittem
  - Research Site, Poederlee
  - Research Site, Poelkapelle
  - Research Site, Quaregnon
  - Research Site, Rance
  - Research Site, Ransart
  - Research Site, Retie
  - Research Site, Retinne
  - Research Site, Roeselare
  - Research Site, Ronse
  - Research Site, Rotheux-Rimière
  - Research Site, Ruiselede
  - Research Site, Saint-Vaast
  - Research Site, Saintes
  - Research Site, Saive
  - Research Site, Schilde
  - Research Site, Selayn
  - Research Site, Sint-Lambrechts-Herk
  - Research Site, Sint-Niklaas
  - Research Site, Staden
  - Research Site, Steenokkerzeel
  - Research Site, Templeuve
  - Research Site, Tessenderlo
  - Research Site, Thuin
  - Research Site, Tielt
  - Research Site, Tubize
  - Research Site, Veurne
  - Research Site, Vosselaar
  - Research Site, Waasmunster
  - Research Site, Wanze
  - Research Site, Waremme
  - Research Site, Wasseiges
  - Research Site, Watervliet
  - Research Site, Wellin
  - Research Site, Wenduine
  - Research Site, Wervik
  - Research Site, Westrozebeke
  - Research Site, Wetteren
  - Research Site, Willebroek
  - Research Site, Wingene
  - Research Site, Zedelgem
  - Research Site, Zemst
  - Research Site, Zoersel
  - Research Site, Zonnebeke
  - Research Site, Zottegem
  - Research Site, Zwevegem
- Greece (29):
  - Research Site, Crete, Crete
  - Research Site, Corfu, Kerkyra
  - Research Site, Lakonia, Lakonia
  - Research Site, Piraeus, Peiraias
  - Research Site, Agrinio
  - Research Site, Alexandroupoli
  - Research Site, Amaliáda
  - Research Site, Arta
  - Research Site, Athens
  - Research Site, Chalcis
  - Research Site, Drama
  - Research Site, Edessa
  - Research Site, Giannitsá
  - Research Site, Grevená
  - Research Site, Ioannina
  - Research Site, Kastoria
  - Research Site, Kavala
  - Research Site, Komotini
  - Research Site, Kos
  - Research Site, Kozani
  - Research Site, Lamia
  - Research Site, Larissa
  - Research Site, Náousa
  - Research Site, Pátrai
  - Research Site, Rhodes
  - Research Site, Serres
  - Research Site, Thessaloniki
  - Research Site, Thérmo
  - Research Site, Volos
- Luxembourg (19):
  - Research Site, Bertrange
  - Research Site, Bissen
  - Research Site, Bridel
  - Research Site, Diekierch
  - Research Site, Differdange
  - Research Site, Dudelange
  - Research Site, Esch-sur-Alzette
  - Research Site, Ettelbruck
  - Research Site, Hollenfels
  - Research Site, Hosingen
  - Research Site, Kehlen
  - Research Site, Larochette
  - Research Site, Luxembourg
  - Research Site, Obercorn
  - Research Site, Redange
  - Research Site, Rodange
  - Research Site, Rumelange
  - Research Site, Sanem
  - Research Site, Strassen
- Portugal (11):
  - Research Site, Beja
  - Research Site, Elvas
  - Research Site, Faro
  - Research Site, Gaia
  - Research Site, Lisbon
  - Research Site, Penafiel
  - Research Site, Porto
  - Research Site, Santarém
  - Research Site, Torres Novas
  - Research Site, Torres Vedras
  - Research Site, Viana do Castelo
- Spain (19):
  - Research Site, Barcelona, Barceloan
  - Research Site, Sant Fruitós de Bages, Barceloan
  - Research Site, Badalona, Barcelona
  - Research Site, Manresa, Barcelona
  - Research Site, Monistrol de Montserrat, Barcelona
  - Research Site, Begonte, Lugo
  - Research Site, Guitiriz, Lugo
  - Research Site, Viveiro, Lugo
  - Research Site, San Fernando de Henares, Madrid
  - Research Site, Ribadesella, Principality of Asturias
  - Research Site, Villar del Arzobispo, Valencia
  - Research Site, Mombuey, Zamora
  - Research Site, Tábara, Zamora
  - Research Site, Letux, Zaragoza
  - Research Site, A Coruña
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Valencia
  - Research Site, Zaragoza
- United Kingdom (24):
  - Research Site, Aldershot
  - Research Site, Atherstone
  - Research Site, Belfast
  - Research Site, Blackburn
  - Research Site, Bolton
  - Research Site, Bradford
  - Research Site, Cardiff
  - Research Site, Coventry
  - Research Site, Crawley
  - Research Site, Crowthorne
  - Research Site, Doncaster
  - Research Site, Glasgow
  - Research Site, Harrow
  - Research Site, High Valleyfield
  - Research Site, Peterborough
  - Research Site, Royal Leamington Spa
  - Research Site, Slough
  - Research Site, Sneinton
  - Research Site, Stevenage
  - Research Site, Sunbury-on-Thames
  - Research Site, Sutton
  - Research Site, Watford
  - Research Site, Wellingborough
  - Research Site, Westbury

REFERENCES:
- [Derived] Tsimihodimos V, Kostapanos MS, Moulis A, Nikas N, Elisaf MS. Effects of benchmarking on the quality of type 2 diabetes care: results of the OPTIMISE (Optimal Type 2 Diabetes Management Including Benchmarking and Standard Treatment) study in Greece. Ther Adv Endocrinol Metab. 2015 Oct;6(5):199-209. doi: 10.1177/2042018815592803. PMID 26445642
- [Derived] Hermans MP, Elisaf M, Michel G, Muls E, Nobels F, Vandenberghe H, Brotons C; OPTIMISE International Steering Committee. Benchmarking is associated with improved quality of care in type 2 diabetes: the OPTIMISE randomized, controlled trial. Diabetes Care. 2013 Nov;36(11):3388-95. doi: 10.2337/dc12-1853. Epub 2013 Jul 11. PMID 23846810
- [Derived] Michel G; OPTIMISE. [The OPTIMISE study (Optimal Type 2 Diabetes Management Including Benchmarking and Standard Treatment]. Results for Luxembourg]. Bull Soc Sci Med Grand Duche Luxemb. 2012;(1):43-9. French. PMID 22822562
- [Derived] Hermans MP, Brotons C, Elisaf M, Michel G, Muls E, Nobels F; (for the OPTIMISE (OPtimal Type 2 dIabetes Management Including benchmarking and Standard trEatment) International Steering Committee). Optimal type 2 diabetes mellitus management: the randomised controlled OPTIMISE benchmarking study: baseline results from six European countries. Eur J Prev Cardiol. 2013 Dec;20(6):1095-105. doi: 10.1177/2047487312449414. Epub 2012 May 17. PMID 22605788
- [Derived] Nobels F, Debacker N, Brotons C, Elisaf M, Hermans MP, Michel G, Muls E; OPTIMISE (OPtimal Type 2 dIabetes Management Including benchmarking and Standard trEatment) International Steering Committee. Study rationale and design of OPTIMISE, a randomised controlled trial on the effect of benchmarking on quality of care in type 2 diabetes mellitus. Cardiovasc Diabetol. 2011 Sep 22;10:82. doi: 10.1186/1475-2840-10-82. PMID 21939502